CLINICAL TRIAL: NCT06189599
Title: Modified Bacteria for Mn-based antioxIdants Production and Delivery for Gut Inflammation Control
Brief Title: Modified antioxIdants Bacteria for Gut Inflammation
Acronym: MOBIDIC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231159
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Chronic Inflammatory Small Bowel Disease
Keywords: IBD; Treatment acceptability; well-being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with IBD experience complex therapeutic pathways. The development of new treatments, more effective and free of side effects, is a therapeutic need. However, such therapeutic innovations can only be effective if they are accepted by the target populations.

The objective of this study is to analyze, in patients with chronic inflammatory bowel diseases, the acceptability of 4 different treatments: chemically modified bacteria treatment, genetically modified bacteria treatment, probiotics, and fecal microbiota transplantation.

The acceptability of the treatments, i.e. the patients' responses and their rationalizations, will constitute the evaluation criterion and the result of the research.

This study will also allow us to evaluate the impact of IBD on quality of life and well-being. Research factors associated with quality of life and well-being, based on dedicated questions (scales validated and included in the questionnaire), evaluate the differential acceptability of the 4 treatments studied. Finally, cross-analyses between health, socio-demographic factors, quality of life and well-being will be performed.

DETAILED DESCRIPTION:
Patients with IBD experience complex treatment pathways. Therapeutic innovations are necessary but can only be effective if they are accepted by the target populations.

It is therefore a question of understanding and measuring the acceptability of innovative treatments for IBD. Through an analysis carried out by the patients regularly followed for a IBD in day hospital will answer questionnaires, to allow us to:

1. understand the representations of competing therapies for this type of pathologies, i.e. conventional drug treatments, probiotics, TMF and CMB and GMB;
2. measure the acceptability of CMB and GMB by the patients themselves;
3. understand the links between the acceptability of treatments and the health status / socio-economic characteristics of patients.

The main criterion for the acceptability of treatments involving bacteria will be the answers to questions relating to this question.

It will be a question of determining which treatment(s) is, or are, the most easily accepted by patients with IBD, understood as a population, understanding why patients prefer this or that treatment, but also "how many" of them say they are ready to use them. In other words, the measures will be based on declarative quantitative questionnaires.

There will be only one interview with each patient, lasting between 15 and 20 minutes.

Recruitment will take place in the gastroenterology and nutrition department of Saint-Antoine Hospital (Paris) and more specifically among patients followed in day hospital and in consultation. This tertiary center has an active queue of 3,300 patients and therefore has the single-center capacity to allow the inclusion of 500 patients for a questionnaire study.

The information notice and the non-objection form will be delivered and collected on the day of the investigation. Once the non-objection has been collected, the questionnaire will be distributed to the patient and then collected before leaving the day hospital.

The collection sheets will be collected in a medical office of the service then entered over time in the dedicated e-CRF (Redcap), before the analysis phase.

The data will be analyzed once the computer entry has been completed in full. The analysis will be done on site by ANR MoBIDIC partners under the supervision of the PI, Philippe SEKSIK. No data or data analysis will be done outside of APHP.

Statistical analyzes will include bivariate and multivariate, parametric and non-parametric analyses. For the latter, binary logistic regressions will be of major use because they will make it possible to determine the factors influencing the acceptability (or rejection) of the treatments studied, taking into account the influence of all these factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic inflammatory bowel diseases.
* Patients over 18 years old.
* Not opposed to participating in the study. - Patients whose diagnosis of IBD was made more than 6 months ago

Exclusion Criteria:

* patients with cognitive disorders,
* patients who cannot read and understand French

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients suffering from IBD and followed in the gastroenterology and nutrition department of Saint-Antoine hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-02-02 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Treatments acceptability | 6 months
  It will be a question of determining which treatment(s) is, or are, the most easily accepted by patients with IBD, understanding why patients prefer this or that treatment, but also "how many" of them say they are ready to use them. In other words, the measures will be based on quantitative declarative questionnaires

SECONDARY OUTCOMES:
Quality of life | 9 months
  Short IBDQ questionnaire (e.g. Williet et al., 2017), cognitive dimension of well-being assessed by the life satisfaction scale (e.g. Duboz et al., 2022, scale validated in French).
Factors associated with quality of life and well-being, based on the questionnaire | 12 months
  Quality of life measured by the short IBDQ questionnaire (e.g. Williet et al., 2017), cognitive dimension of well-being assessed by the life satisfaction scale (e.g. Duboz et al., 2022, scale validated in French).
  Research into factors associated with quality of life and well-being, based on the questionnaire: bivariate and multivariate analyses.
Differential acceptability of the 4 treatments studied | 12 months
  Comparison of acceptability rates using Chi2 tests. Cross-analyses between health indicators, socio-demographic factors, quality of life and well-being: based on the questionnaires, dedicated statistical analyses (correlations, Student tests, ANOVA, Chi2, regressions, cluster analyses).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Seksik, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Gastroentérologie en Nutrition - Hôpital St Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No
Data will be collected and analyzed on site